CLINICAL TRIAL: NCT01528657
Title: Ventricular Pace Suppression Versus Intrinsic Rhythm Support Study
Acronym: VIPERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA098
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Sick Sinus Syndrome
Keywords: Sick Sinus Syndrome; Ventricular pacing; Minimal ventricular pacing; Ventricular pacing suppression; Intrinsic rhythm support; Long term AV
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ventricular Pace Suppression (VpS) (Experimental): The function Ventricular Pace Suppression (VpS) is activated
  Interventions: Other: Ventricular Pace Suppression (Vps)
- Intrinsic Rhythm Support (IRSplus) (Experimental): The function Intrinsic Rhythm Support (IRSplus) is activated
  Interventions: Other: Intrinsic rhythm support (IRSplus)

INTERVENTIONS:
Other: Ventricular Pace Suppression (Vps) — Unnecessary ventricular pacing is avoided by promoting intrinsic conduction. In case of intrinsic conduction, the device switches from a DDD mode to an ADI mode.
  Arms: Ventricular Pace Suppression (VpS)
Other: Intrinsic rhythm support (IRSplus) — All parameters of the AV hysteresis functions are set in a way to maintain spontaneous AV conduction of the patient's heart as long as possible.
  Arms: Intrinsic Rhythm Support (IRSplus)

SUMMARY:
The objective of this study is to intra-individually compare the performances of two pacemaker algorithms designed to reduce unnecessary right ventricular pacing: Intrinsic Rhythm Support Plus (IRSplus) and Ventricular Pace Suppression (VpS). The study will compare ventricular pacing percentage, long-term atrio-ventricular conduction time, occurrences of atrial tachyarrhythmic events and atrial fibrillation burden percentage in patients implanted with a pacemaker for Sick Sinus Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age;
* Patient has proven informed consent;
* Subject with indication of dual chamber pacemaker due to Sinus Node Dysfunction;
* Subjects with a dual chamber pacemaker already implanted within six months from enrollment, provided that ventricular pacing percentage ≤ 40% and with the right ventricular lead in the apical position;
* Stable medical situation;
* Stable geographical situation;

Exclusion Criteria:

* Permanent or paroxysmal AV block ≥ II;
* Permanent Atrial fibrillation/Atrial flutter;
* Device Replacement;
* Patient with a poor echocardiographic window;
* Patient already implanted with the right ventricular lead not in the apical position;
* Subjects with a dual chamber pacemaker, implanted later than six months;
* Subjects with a dual chamber pacemaker with ventricular pacing percentage ≥ 40%;
* Contraindication for DDD(R)-ADI(R) or DDD(R) pacing modes;
* VpS or IRSplus algorithm contraindications;
* Age < 18 years;
* Life expectancy < 12 months;
* Cardiac surgery planned within the FU period;
* Participation to another clinical investigation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2011-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Ventricular pacing percentage | 6 months

SECONDARY OUTCOMES:
Long-term atrio-ventricular conduction delay | 6 Months
Occurrence of atrial tachycardia or atrial fibrillation events | 6 Months
Burden of atrial fibrillation | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Capucci, Principal Investigator — A.O.U. Ospedali Riuniti, Ancona; Valeria Calvi, Principal Investigator — A.O.U. Policlinico-Vittorio Emanuele, Catania; Marco Brieda, Principal Investigator — A.O. Santa Maria degli Angeli, Pordenone; Ennio Pisanò, Principal Investigator — P.O. Vito Fazzi, Lecce; Vittorio Giudici, Principal Investigator — Ospedale Bolognini, Seriate
Locations (20):
- Italy (20):
  - Ospedale Bolognini, Seriate, Bergamo
  - P.O. F. Ferrari, Casarano, Lecce
  - A.O. Destra Secchia, Pieve di Coriano, Mantova
  - Ospedale San Leonardo, Castellammare di Stabia, Napoli
  - Ospedale SS. Trinità, Borgomanero, Novara
  - Ospedale SS. Cosma e Damiano, Pescia, Pistoia
  - Ospedale Santa Croce, Moncalieri, Torino
  - Ospedale S.Antonio Abate, Gallarate, Varese
  - Ospedale Dell'Angelo, Mestre, Venezia
  - A.O.U. Ospedali Riuniti di Ancona, Ancona
  - Ospedale Degli Infermi, Biella
  - A.O.U. Policlinico-Vittorio Emanuele, Catania
  - Ospedale S. Giuseppe, Empoli
  - Osp. Civile F. Veneziale, Isernia
  - P.O. Vito Fazzi, Lecce
  - A.O.R.N. dei Colli - PO "V. Monaldi", Napoli
  - A.O. Santa Maria Degli Angeli, Pordenone
  - A.O. San Carlo, Potenza
  - Ospedale Degli Infermi, Rimini
  - Ospedale SS. Giovanni e Paolo, Venezia

REFERENCES:
- [Background] Vassallo JA, Cassidy DM, Miller JM, Buxton AE, Marchlinski FE, Josephson ME. Left ventricular endocardial activation during right ventricular pacing: effect of underlying heart disease. J Am Coll Cardiol. 1986 Jun;7(6):1228-33. doi: 10.1016/s0735-1097(86)80140-1. PMID 3711479
- [Background] Prinzen FW, Peschar M. Relation between the pacing induced sequence of activation and left ventricular pump function in animals. Pacing Clin Electrophysiol. 2002 Apr;25(4 Pt 1):484-98. doi: 10.1046/j.1460-9592.2002.00484.x. PMID 11991375
- [Background] Prinzen FW, Augustijn CH, Arts T, Allessie MA, Reneman RS. Redistribution of myocardial fiber strain and blood flow by asynchronous activation. Am J Physiol. 1990 Aug;259(2 Pt 2):H300-8. doi: 10.1152/ajpheart.1990.259.2.H300. PMID 2386214
- [Background] Thambo JB, Bordachar P, Garrigue S, Lafitte S, Sanders P, Reuter S, Girardot R, Crepin D, Reant P, Roudaut R, Jais P, Haissaguerre M, Clementy J, Jimenez M. Detrimental ventricular remodeling in patients with congenital complete heart block and chronic right ventricular apical pacing. Circulation. 2004 Dec 21;110(25):3766-72. doi: 10.1161/01.CIR.0000150336.86033.8D. Epub 2004 Dec 6. PMID 15583083
- [Background] Kanzaki H, Bazaz R, Schwartzman D, Dohi K, Sade LE, Gorcsan J 3rd. A mechanism for immediate reduction in mitral regurgitation after cardiac resynchronization therapy: insights from mechanical activation strain mapping. J Am Coll Cardiol. 2004 Oct 19;44(8):1619-25. doi: 10.1016/j.jacc.2004.07.036. PMID 15489094
- [Background] Maurer G, Torres MA, Corday E, Haendchen RV, Meerbaum S. Two-dimensional echocardiographic contrast assessment of pacing-induced mitral regurgitation: relation to altered regional left ventricular function. J Am Coll Cardiol. 1984 Apr;3(4):986-91. doi: 10.1016/s0735-1097(84)80357-5. PMID 6707363
- [Background] Vanderheyden M, Goethals M, Anguera I, Nellens P, Andries E, Brugada J, Brugada P. Hemodynamic deterioration following radiofrequency ablation of the atrioventricular conduction system. Pacing Clin Electrophysiol. 1997 Oct;20(10 Pt 1):2422-8. doi: 10.1111/j.1540-8159.1997.tb06081.x. PMID 9358483
- [Background] Nielsen JC, Kristensen L, Andersen HR, Mortensen PT, Pedersen OL, Pedersen AK. A randomized comparison of atrial and dual-chamber pacing in 177 consecutive patients with sick sinus syndrome: echocardiographic and clinical outcome. J Am Coll Cardiol. 2003 Aug 20;42(4):614-23. doi: 10.1016/s0735-1097(03)00757-5. PMID 12932590
- [Background] Nielsen JC, Andersen HR, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Heart failure and echocardiographic changes during long-term follow-up of patients with sick sinus syndrome randomized to single-chamber atrial or ventricular pacing. Circulation. 1998 Mar 17;97(10):987-95. doi: 10.1161/01.cir.97.10.987. PMID 9529267
- [Background] Nahlawi M, Waligora M, Spies SM, Bonow RO, Kadish AH, Goldberger JJ. Left ventricular function during and after right ventricular pacing. J Am Coll Cardiol. 2004 Nov 2;44(9):1883-8. doi: 10.1016/j.jacc.2004.06.074. PMID 15519023
- [Background] Sweeney MO, Hellkamp AS, Ellenbogen KA, Greenspon AJ, Freedman RA, Lee KL, Lamas GA; MOde Selection Trial Investigators. Adverse effect of ventricular pacing on heart failure and atrial fibrillation among patients with normal baseline QRS duration in a clinical trial of pacemaker therapy for sinus node dysfunction. Circulation. 2003 Jun 17;107(23):2932-7. doi: 10.1161/01.CIR.0000072769.17295.B1. Epub 2003 Jun 2. PMID 12782566
- [Derived] Calvi V, Pisano EC, Brieda M, Melissano D, Castaldi B, Guastaferro C, Nigro G, Madalosso M, Orsida D, Rovai N, Gargaro A, Capucci A. Atrioventricular Interval Extension Is Highly Efficient in Preventing Unnecessary Right Ventricular Pacing in Sinus Node Disease: A Randomized Cross-Over Study Versus Dual- to Atrial Single-Chamber Mode Switch. JACC Clin Electrophysiol. 2017 May;3(5):482-490. doi: 10.1016/j.jacep.2016.11.011. Epub 2017 Feb 1. PMID 29759604